CLINICAL TRIAL: NCT00517920
Title: An Open-Label, Phase 2 Study of Efficacy and Tolerability of ABT-869 in Advanced Hepatocellular Carcinoma (HCC)
Brief Title: Phase 2 Study of ABT-869 in Advanced Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M06-879
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Advanced Hepatocellular Carcinoma
MeSH Terms: interventions — linifanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABT-869 (Experimental)
  Interventions: Drug: ABT-869

INTERVENTIONS:
Drug: ABT-869 — 0.25 mg/kg QD

SUMMARY:
Phase 2 Study of ABT-869 in Advanced Hepatocellular Carcinoma (HCC)

DETAILED DESCRIPTION:
An Open-label, Phase 2 study of efficacy and tolerability of ABT-869 in advanced hepatocellular carcinoma (HCC)

ELIGIBILITY:
Inclusion Criteria

* Subject must be greater than or equal to 18 years of age
* Subject must be diagnosed with unresectable or metastatic HCC
* Subjects must have a measurable lesion by RECIST on CT scan in at least one site which has not received radiation
* Subject has an Eastern Cooperative Oncology Group (ECOG) Performance status of 0-2
* No other active malignancy within the past 5 years

Exclusion Criteria

* Subject has received targeted VEGF/PDGF/TKI therapy. Prior Avastin is allowed
* Subject has Child-Pugh grade Class C hepatic impairment
* The subject has proteinuria Common Toxicity Criteria (CTC) grade > 1 as measured by routine urinalysis or 24 hour urine collection during screening assessment
* Subject currently exhibits symptomatic or persistent, uncontrolled hypertension defined as diastolic blood pressure > 100 mmHg or systolic blood pressure > 150 mmHg. Subjects may be re-screened if blood pressure is shown to be controlled with or without intervention
* The subject has a documented left ventricular Ejection Fraction < 50%
* Subject is receiving therapeutic anticoagulation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-09; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Progression-Free Rate | Week 16
Objective Response Rate | Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Justin Ricker, MD, Study Director — AbbVie
Locations (6):
- Site Reference ID/Investigator# 7726, Philadelphia, Pennsylvania, United States
- Canada (2):
  - Site Reference ID/Investigator# 7169, Toronto
  - Site Reference ID/Investigator# 5837, Vancouver
- Singapore (2):
  - Site Reference ID/Investigator# 5235, Singapore
  - Site Reference ID/Investigator# 5611, Singapore
- Site Reference ID/Investigator# 6265, Taipei, Taiwan